CLINICAL TRIAL: NCT00463151
Title: An Exploratory Study of Rebamipide in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Saito Katsuhisa, OPCJ
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 037-06-001; JapicCTI-070399 (Other: Japic)
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Colitis, Ulcerative
Keywords: Rebamipide; Enema; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): 0mg rebamipide
  Interventions: Drug: rebamipide
- 2 (Experimental): 60mg rebamipide
  Interventions: Drug: rebamipide
- 3 (Experimental): 150mg rebamipide
  Interventions: Drug: rebamipide
- 4 (Experimental): 300mg rebamipide
  Interventions: Drug: rebamipide

INTERVENTIONS:
Drug: rebamipide — 0, 60, 150, 300mg of rebamipide per day for 6 weeks into colon

SUMMARY:
The purpose of this study is to examine the safety and efficacy of rebamipide by once daily intracolonial administration at 0 (placebo), 60, 150, or 300 mg for 6 weeks in patients with active ulcerative colitis, who are being treated with oral aminosalicylic acid (ASA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active ulcerative colitis
2. Patients having an insufficient response to ASA oral formulation: (1) Patients whose ongoing use of ASA oral formulation from ≥2 weeks prior to the day before registration is fixed at mesalazine ≥2 g/day or salazosulfapyridine 3-6 g/day, (2) Patients with continuous bloody stools from ≥2 weeks prior to the day before registration, (3) Patients whose DAI subscores are ≥2 points for "bloody stools" and ≥2 points for "endoscopic findings"
3. Patients shown via colonoscopy to have major lesions between the sigmoid colon and rectum (with lesions not extending beyond the splenic flexure)
4. Outpatients

Exclusion Criteria:

1. Patients who have a history of intestinal resection (other than appendiceal resection)
2. Patients who have a complication of malignant tumor
3. Female patients who are pregnant, lactating, or possibly pregnant, or who hope to become pregnant during the study period
4. Patients who have complications of serious cardiac, hepatic or renal impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (5):
- Japan (5):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kinki Region
  - Kyushu Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebamipide 60 mg: Once daily intracolonial administration at a dose of 60 mg for 6 weeks
- Rebamipide 150 mg: Once daily intracolonial administration at a dose of 150 mg for 6 weeks
- Rebamipide 300 mg: Once daily intracolonial administration at a dose of 300 mg for 6 weeks
- Placebo: Once daily intracolonial administration of placebo for 6 weeks
Period: Overall Study
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
Started | 35 | 29 | 29 | 31
Completed | 33 | 24 | 26 | 24
Not Completed | 2 | 5 | 3 | 7
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 5 | 2 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: subjects who received at least one dose of the study drug and for whom postdose efficacy data were obtained
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo | Total
Number analyzed (Participants) | 35 | 29 | 27 | 30 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 26 | 25 | 28 | 113
  >=65 years | 1 | 3 | 2 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 8 | 14 | 52
  Male | 21 | 13 | 19 | 16 | 69
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 35 | 29 | 27 | 30 | 121

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement Rate (Number of Subjects Showing Clinical Improvement/Number of Subjects Evaluated x 100)
Description: Definition of clinical improvement: a decrease of Disease Activity Index [DAI] score for "rectal bleeding" to either 0 or 1 point and a decrease of ≥1 point in the DAI score for "findings on endoscopy" from the baseline
Time Frame: Week 6
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
Number analyzed (Participants) | 35 | 29 | 27 | 30
percentage of participants | 31.4 [16.0 to 46.8] | 24.1 [8.6 to 39.7] | 44.4 [25.7 to 63.2] | 30.0 [13.6 to 46.4]

2. Secondary Outcome: Clinical Remission (Number of Subjects Showing Remission/Number of Subjects Evaluated x 100)
Description: Definition of remission: a decrease of the total DAI scores for "rectal bleeding" and "findings on endoscopy" to 0 points
Time Frame: Week 6
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
Number analyzed (Participants) | 35 | 29 | 27 | 30
percentage of participants | 2.9 [0.0 to 8.4] | 0.0 [0.0 to 0.0] | 18.5 [3.9 to 33.2] | 3.3 [0.0 to 9.8]

3. Secondary Outcome: Mean Change From Baseline in Total DAI Score
Description: DAI measures disease activity through assessment of 4 items/subscales: stool frequency, rectal bleeding, findings on endoscopy, and physician's global assessment. Each item of the score is assessed on a 4-point scale from 0 to 3; the total score ranges from 0 to 12 with a higher score representing greater severity. A negative change in mean score indicates improvement.
Time Frame: Baseline and Week 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
Number analyzed (Participants) | 33 | 26 | 26 | 27
score on a scale | -2.5 (2.5) | -1.6 (2.6) | -3.0 (3.0) | -2.0 (2.1)

4. Secondary Outcome: Percentage of Subjects Showing Improvement in Each DAI Subscore
Description: DAI measures disease activity through assessment of 4 items/subscales: stool frequency, rectal bleeding, findings on endoscopy, and physician's global assessment. Each item of the score is assessed on a 4-point scale from 0 to 3 with a higher score representing greater severity. A negative change from baseline indicates improvement.
Time Frame: Baseline and week 6
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
Number analyzed (Participants) | 35 | 29 | 27 | 30
percentage of participants
  Stool frequency | 48.6 | 31.0 | 59.3 | 10.0
  Rectal bleeding | 65.7 | 51.7 | 66.7 | 63.3
  Findings on endoscopy: number analyzed (Participants) | 33 | 26 | 26 | 27
  Findings on endoscopy | 39.4 | 26.9 | 53.8 | 48.1
  Physician's global assessment | 48.6 | 31.0 | 51.9 | 36.70

5. Secondary Outcome: Mean Change From Baseline in Total Endoscopic Index (EI) Score
Description: The index consisted of 4 subscales: granulation scattering reflected light, vascular pattern, vulnerability of mucosa, and mucosal damage. Each subscale was scored on a scale of 0 to 4 and the total score (the sum of all 4 subscores) ranges from 0 to 12, higher scores indicate more severe disease.
Time Frame: Baseline and Week 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
Number analyzed (Participants) | 33 | 26 | 26 | 27
score on a scale | -1.6 (2.2) | -1.2 (2.5) | -2.4 (2.9) | -1.9 (2.4)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Day 1 (start of treatment) up to approximately 10 weeks
Description: Safety Set comprised subjects who received the study drug at least once.
Arm/Group | Rebamipide 60 mg | Rebamipide 150 mg | Rebamipide 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/29 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/35 | 2/29 | 0/29 | 1/31
Other Adverse Events (participants affected / at risk) | 22/35 | 20/29 | 18/29 | 22/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebamipide 60 mg (N=35) | Rebamipide 150 mg (N=29) | Rebamipide 300 mg (N=29) | Placebo (N=31)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebamipide 60 mg (N=35) | Rebamipide 150 mg (N=29) | Rebamipide 300 mg (N=29) | Placebo (N=31)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 2 | 6 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 3 | 1 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Basophil count increased (Investigations) | 0 | 2 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 2
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 2
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 2 | 1 | 2
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 2 | 0 | 1 | 1
Eosinophil count decreased (Investigations) | 0 | 0 | 1 | 1
Eosinophil count increased (Investigations) | 1 | 3 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 0
Glucose urine present (Investigations) | 1 | 1 | 1 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count abnormal (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Monocyte count increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Red blood cell count increased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1
White blood cell count increased (Investigations) | 3 | 3 | 0 | 4
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 2 | 2 | 1 | 2
Protein urine present (Investigations) | 1 | 2 | 1 | 1
Urine ketone body present (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 3 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No